CLINICAL TRIAL: NCT02860130
Title: Clinical Evaluation of Use of Prismocitrate 18 in Patients Undergoing Acute Continuous Renal Replacement Therapy (CRRT)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study halted due to low recruitment, unrelated to safety or efficacy reasons
Sponsor: Vantive Health LLC (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1407-004
Record Dates: First submitted 2016-07-29; First posted 2016-08-09 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Regional Citrate Anticoagulation (RCA); Continuous Renal Replacement Therapy (CRRT); Acute Kidney Injury
Keywords: Regional Citrate Anticoagulation (RCA); Continuous Renal Replacement Therapy (CRRT); Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prismocitrate 18 (Experimental)
  Interventions: Drug: Prismocitrate 18
- No Regional Anticoagulation of CRRT Circuit (Active Comparator)
  Interventions: Other: No Anticoagulation

INTERVENTIONS:
Drug: Prismocitrate 18 — Modality of CVVHDF
  Other Names: Regional Citrate Anticoagulation (RCA)
  Arms: Prismocitrate 18
Other: No Anticoagulation — Modality of CVVHDF
  Arms: No Regional Anticoagulation of CRRT Circuit

SUMMARY:
The purpose of this research is to determine if an investigational new drug solution called Prismocitrate 18 lengthens extracorporeal circuit life in patients treated with continuous renal replacement therapy (CRRT). Patients who receive CRRT treatment with Prismocitrate 18 as the anticoagulant will be compared to patients who receive CRRT treatment with no anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be receiving medical care in an intensive care unit (ICU) (e.g., medical ICU, surgical ICU, cardiothoracic ICU, Trauma ICU, Mixed ICU, other).
2. Adult patients with AKI or other serious conditions who require treatment with CRRT.
3. Patients are expected to remain in the ICU and on CRRT for at least 72 hours after randomization.
4. Patients already receiving standard-of-care CRRT must be randomized within 24 hours of initiation of their standard-of-care CRRT.

Exclusion Criteria:

1. Patients requiring systemic anticoagulation with antithrombotic agents for reasons other than CRRT. The exception is patients receiving subcutaneous heparin for deep vein thrombosis prophylaxis according to institutional practice or patients on aspirin may be enrolled.
2. Patients in whom citrate anticoagulation is contraindicated such as patients with a known allergy to citrate or who have experienced adverse events associated with citrate products including patients with a prior history of citrate toxicity or patients with uncorrected severe hypocalcemia (whether in the context of current citrate administration or due to the underlying disease state).
3. Patients who are not candidates for CRRT.
4. Patients who are receiving extracorporeal membrane oxygenation (ECMO) therapy.
5. Patients with severe coagulopathy [i.e., platelets < 30,000/mm3, international normalized ratio (INR) > 2, partial thromboplastin time (PTT) > 50 seconds] including severe thrombocytopenia (platelets < 30,000/mm3), HIT (heparin induced thrombocytopenia), ITP (idiopathic thrombocytopenia purpura), and TTP (thrombotic thrombocytopenia purpura) should not be enrolled in the trial.
6. Patients with fulminant acute liver failure or acute on chronic liver failure as documented by a Child-Pugh Liver Failure Score > 10.
7. Patients with refractory shock associated persistent, worsening with lactic acidosis (lactate > 4 mmol/L). However, patients with improving subsequent serum lactate levels may be enrolled.
8. Patients unlikely to survive at least 72 hours.
9. Female patients who are pregnant, lactating, or planning to become pregnant during the study period.
10. Patients who are currently participating in another interventional clinical study.
11. Patients with a medical condition that may interfere with the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2018-05-12 (Actual); Study Completion 2018-05-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Beth Israel Deaconess (Harvard), Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cleveland Clinic, Cleveland, Ohio
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tsujimoto H, Tsujimoto Y, Nakata Y, Fujii T, Takahashi S, Akazawa M, Kataoka Y. Pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2020 Dec 14;12(12):CD012467. doi: 10.1002/14651858.CD012467.pub3. PMID 33314078

RESULTS

PARTICIPANT FLOW:
Groups:
- Prismocitrate 18: CRRT with Prismocitrate 18 solution. If a patient was already receiving standard-of-care CRRT, they were required to be randomized within 24 hours of initiation of their standard-of-care CRRT. All patients were treated with pre-dilution CVVHDF as the study CRRT modality. Extracorporeal circuit life was monitored for up to 120 hours of study CRRT (Treatment Period).
- No Systemic Anticoagulation: CRRT with no systemic anticoagulation. If a patient was already receiving standard-of-care CRRT, they were required to be randomized within 24 hours of initiation of their standard-of-care CRRT. All patients were treated with pre-dilution CVVHDF as the study CRRT modality. Extracorporeal circuit life was monitored for up to 120 hours of study CRRT (Treatment Period).
Period: Overall Study
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Started | 17 | 17
Completed | 10 | 8
Not Completed | 7 | 9
Not completed — Adverse Event | 2 | 3
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Physician Decision | 2 | 2
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Population: FAS
Groups:
- Total: Total of all reporting groups
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Customized [Count of Participants; unit: Participants]
  ≥ 18 years to ≤ 35 years | 1 | 0 | 1
  > 35 years to ≤ 45 years | 2 | 1 | 3
  > 45 years to ≤ 55 years | 1 | 3 | 4
  > 55 years to ≤ 65 years | 4 | 4 | 8
  > 65 years | 9 | 9 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 11 | 7 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 8 | 10
  White | 15 | 9 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Time to Occurrence of Selected Prismaflex® System Alarms/Conditions
Description: The point estimate is time point (number of hours of the extracorporeal circuit life of a filter) at which (100-percentile)% filters are still surviving (i.e. number surviving divided by number at risk), based on the Kaplan-Meier method. For example, for the 25th percentile: after 33.18 hours, 75% of filters are still surviving. Given the early termination, this study was not powered to show statistically significant changes in efficacy endpoints. The Prismaflex M150 Set extracorporeal circuit life of filters were intended to be assessed over a maximum of 120 hours (Treatment Period) by duration of time for which each Prismaflex M150 Set could be used continuously over a maximum 72 hour time-period in each patient. The end of the extracorporeal circuit life was defined by the occurrence of one or both of the following Prismaflex® System alarms/conditions if the alarms could not be mitigated: (1) "Warning: Filter Clotted", and/or (2) "Advisory transmembrane pressure (TMP) Too High."
Time Frame: Up to 120 hours post CRRT treatment initiation
Population: Full Analysis Set (FAS)-randomized treatment groups (intent-to-treat principle)
Measure: Number (95% Confidence Interval); unit: hours
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
hours
  25 Percentile | 33.180 [8.340 to NA] — Not reached due to early termination of study. | 17.680 [11.990 to 24.070]
  50 Percentile | NA [NA to NA] — Not reached due to early termination of study. | 29.660 [23.730 to NA] — Not reached due to early termination of study.
  75 Percentile | NA [NA to NA] — Not reached due to early termination of study. | NA [32.500 to NA] — Not reached due to early termination of study.

2. Secondary Outcome: Change From Baseline in Patient Ionized Calcium (iCa) by Hour
Description: Systemic blood iCa concentrations
Time Frame: Baseline and up to 120 hours post CRRT treatment initiation
Population: Overall Number of Participants Analyzed (N) reflects FAS, and number of subjects (n) with evaluable data is shown for each individual timepoint.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
mmol/L
  1 Hour: number analyzed (Participants) | 13 | 15
  1 Hour | -0.1 (0.14) | 0 (0.06)
  6 Hours: number analyzed (Participants) | 14 | 16
  6 Hours | -0.1 (0.11) | 0 (0.07)
  12 Hours: number analyzed (Participants) | 13 | 16
  12 Hours | -0.0 (0.17) | 0 (0.1)
  18 Hours: number analyzed (Participants) | 14 | 16
  18 Hours | 0 (0.18) | 0 (0.12)
  24 Hours: number analyzed (Participants) | 12 | 16
  24 Hours | 0.1 (0.19) | -0.0 (0.17)
  30 Hours: number analyzed (Participants) | 12 | 13
  30 Hours | 0 (0.17) | 0 (0.13)
  36 Hours: number analyzed (Participants) | 13 | 13
  36 Hours | 0 (0.14) | -0.0 (0.12)
  42 Hours: number analyzed (Participants) | 13 | 13
  42 Hours | 0 (0.18) | 0 (0.15)
  48 Hours: number analyzed (Participants) | 13 | 13
  48 Hours | 0 (0.15) | 0 (0.16)
  54 hours: number analyzed (Participants) | 13 | 12
  54 hours | 0 (0.14) | -0.0 (0.15)
  60 hours: number analyzed (Participants) | 12 | 11
  60 hours | 0 (0.12) | -0.0 (0.15)
  66 Hours: number analyzed (Participants) | 13 | 12
  66 Hours | -0.0 (0.14) | -0.0 (0.15)
  72 Hours: number analyzed (Participants) | 13 | 11
  72 Hours | 0 (0.13) | 0 (0.16)
  78 Hours: number analyzed (Participants) | 11 | 10
  78 Hours | 0 (0.16) | 0 (0.16)
  84 Hours: number analyzed (Participants) | 11 | 9
  84 Hours | 0 (0.15) | -0.0 (0.17)
  90 Hours: number analyzed (Participants) | 11 | 9
  90 Hours | 0 (0.17) | -0.0 (0.15)
  96 Hours: number analyzed (Participants) | 11 | 9
  96 Hours | 0 (0.11) | -0.0 (0.16)
  102 Hours: number analyzed (Participants) | 11 | 8
  102 Hours | 0 (0.14) | 0 (0.16)
  108 Hours: number analyzed (Participants) | 11 | 7
  108 Hours | 0 (0.14) | 0 (0.16)
  114 Hours: number analyzed (Participants) | 9 | 7
  114 Hours | 0.1 (0.13) | 0 (0.15)
  120 Hours: number analyzed (Participants) | 7 | 6
  120 Hours | 0.1 (0.14) | -0.0 (0.15)

3. Secondary Outcome: Extracorporeal Circuit Ionized Calcium by Hour
Description: Post-filter blood iCa concentrations will only be measured in the Prismocitrate 18 arm. The extracorporeal circuit (post-filter).
Time Frame: Up to 120 hours post CRRT treatment initiation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Prismocitrate 18
Number analyzed (Participants) | 17
mmol/L
  1 Hour: number analyzed (Participants) | 16
  1 Hour | 0.5 (0.11)
  6 Hours: number analyzed (Participants) | 14
  6 Hours | 0.5 (0.13)
  12 Hours: number analyzed (Participants) | 14
  12 Hours | 0.5 (0.11)
  18 Hours: number analyzed (Participants) | 16
  18 Hours | 0.5 (0.11)
  24 Hours: number analyzed (Participants) | 14
  24 Hours | 0.5 (0.11)
  30 Hours: number analyzed (Participants) | 15
  30 Hours | 0.5 (0.11)
  36 Hours: number analyzed (Participants) | 15
  36 Hours | 0.5 (0.1)
  42 Hours: number analyzed (Participants) | 14
  42 Hours | 0.5 (0.23)
  48 Hours: number analyzed (Participants) | 13
  48 Hours | 0.5 (0.12)
  54 hours: number analyzed (Participants) | 14
  54 hours | 0.5 (0.11)
  60 hours: number analyzed (Participants) | 13
  60 hours | 0.5 (0.13)
  66 Hours: number analyzed (Participants) | 14
  66 Hours | 0.5 (0.17)
  72 Hours: number analyzed (Participants) | 14
  72 Hours | 0.4 (0.1)
  78 Hours: number analyzed (Participants) | 13
  78 Hours | 0.4 (0.12)
  84 Hours: number analyzed (Participants) | 13
  84 Hours | 0.4 (0.11)
  90 Hours: number analyzed (Participants) | 11
  90 Hours | 0.4 (0.1)
  96 Hours: number analyzed (Participants) | 12
  96 Hours | 0.4 (0.11)
  102 Hours: number analyzed (Participants) | 12
  102 Hours | 0.4 (0.13)
  108 Hours: number analyzed (Participants) | 12
  108 Hours | 0.4 (0.11)
  114 Hours: number analyzed (Participants) | 10
  114 Hours | 0.4 (0.11)
  120 Hours: number analyzed (Participants) | 7
  120 Hours | 0.5 (0.16)

4. Secondary Outcome: Delivery of Prescribed CRRT Dose by Day
Description: Evaluates the efficacy of using Prismocitrate 18 in delivering the prescribed CRRT dose, with delivered dose based on (daily) average effluent rate divided by (daily) average weight and expressed as mL/kg/hour.
Time Frame: Up to 120 hours post CRRT treatment initiation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/kg/hour
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
mL/kg/hour
  Day 1: number analyzed (Participants) | 16 | 16
  Day 1 | 32.3 (7.064) | 30.34 (7.407)
  Day 2: number analyzed (Participants) | 13 | 13
  Day 2 | 33.12 (9.676) | 32.49 (10.191)
  Day 3: number analyzed (Participants) | 11 | 11
  Day 3 | 31.62 (8.045) | 32.29 (10.533)
  Day 4: number analyzed (Participants) | 8 | 8
  Day 4 | 31.93 (10.187) | 35.19 (10.95)
  Day 5: number analyzed (Participants) | 8 | 8
  Day 5 | 32.83 (11.119) | 33.31 (13.103)

5. Secondary Outcome: Number of Investigator Site Facilities That Passed Prismocitrate 18 Training Assessment
Description: Training conducted on administration of Prismocitrate 18 to demonstrate the understanding of the user groups on how to use the solution by passing an assessment at the end of training. The user groups who needed to be assessed prior to use of Prismocitrate 18 in the clinical trial setting were to be comprised of physicians, nurses, and other clinicians who were part of prescribing, initiating or modifying treatment during the 120 hour Treatment Period. The training assessment was housed on a restricted access study website. Study personnel who completed the training assessment have a completion date listed which indicates that the individual received a passing score of 80% or better on the training assessment.
Time Frame: Prior to study use of Prismocitrate 18
Population: Physicians, nurses, and other clinicians who were part of prescribing, initiating or modifying treatment at each Investigator site. Staff at each site facility passed testing, but the overall number of participants is not known. No analysis of investigator training test scores were conducted as results for individual test questions were not retained for analysis.
Measure: Number; unit: site facility staff
Units Other Than Participants: site facilities
Arm/Group | Prismocitrate 18
Number analyzed (Participants) | NA
Number analyzed (site facilities) | 6
site facility staff | 6

6. Secondary Outcome: Change From Baseline in Serum Bicarbonate by Hour
Time Frame: Baseline and up to 120 hours post CRRT treatment initiation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
mmol/L
  6 Hours: number analyzed (Participants) | 12 | 13
  6 Hours | 0.2 (3.86) | 2.4 (3.48)
  12 Hours: number analyzed (Participants) | 14 | 15
  12 Hours | 0.8 (4.42) | 2.9 (3.27)
  18 Hours: number analyzed (Participants) | 15 | 16
  18 Hours | 1.3 (5.43) | 2.3 (4.11)
  24 Hours: number analyzed (Participants) | 16 | 14
  24 Hours | 2.8 (4.64) | 2 (4.99)
  30 Hours: number analyzed (Participants) | 15 | 13
  30 Hours | 2.9 (5.02) | 2.9 (4.21)
  36 Hours: number analyzed (Participants) | 16 | 12
  36 Hours | 3.3 (5.6) | 2.6 (3.71)
  42 Hours: number analyzed (Participants) | 16 | 12
  42 Hours | 3.3 (5.52) | 3.6 (3.61)
  48 Hours: number analyzed (Participants) | 15 | 13
  48 Hours | 2.7 (5.56) | 2.4 (3.99)
  54 Hours: number analyzed (Participants) | 14 | 10
  54 Hours | 2.7 (5.72) | 2.1 (3.77)
  60 Hours: number analyzed (Participants) | 13 | 11
  60 Hours | 4.7 (6.56) | 2.4 (4.29)
  66 Hours: number analyzed (Participants) | 15 | 8
  66 Hours | 3.7 (6.49) | 2.6 (5.02)
  72 Hours: number analyzed (Participants) | 16 | 10
  72 Hours | 4.2 (6.59) | 0.1 (6.68)
  78 Hours: number analyzed (Participants) | 13 | 8
  78 Hours | 2.8 (5.01) | 2.9 (5.46)
  84 Hours: number analyzed (Participants) | 13 | 9
  84 Hours | 3.3 (5.48) | 2.5 (5.34)
  90 Hours: number analyzed (Participants) | 12 | 8
  90 Hours | 3.3 (6.05) | 2.2 (5.26)
  96 Hours: number analyzed (Participants) | 12 | 8
  96 Hours | 2.8 (5.88) | 1.4 (5.81)
  102 Hours: number analyzed (Participants) | 11 | 5
  102 Hours | 2.2 (5.64) | -1.1 (7.48)
  108 Hours: number analyzed (Participants) | 12 | 7
  108 Hours | 2.7 (5.25) | -0.4 (7.67)
  114 Hours: number analyzed (Participants) | 10 | 5
  114 Hours | 3.8 (6.2) | -2.8 (8)
  120 Hours: number analyzed (Participants) | 8 | 6
  120 Hours | 2.8 (5.94) | -1.5 (7.13)

7. Secondary Outcome: Change From Baseline in pH by Hour
Time Frame: Baseline and up to 120 hours post CRRT treatment initiation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
pH
  6 Hours: number analyzed (Participants) | 12 | 13
  6 Hours | -0.0 (0.06) | 0.1 (0.09)
  12 Hours: number analyzed (Participants) | 13 | 15
  12 Hours | -0.0 (0.07) | 0.1 (0.1)
  18 Hours: number analyzed (Participants) | 15 | 15
  18 Hours | 0 (0.1) | 0 (0.11)
  24 Hours: number analyzed (Participants) | 16 | 14
  24 Hours | 0 (0.1) | 0 (0.1)
  30 Hours: number analyzed (Participants) | 14 | 10
  30 Hours | 0 (0.1) | 0.1 (0.11)
  36 Hours: number analyzed (Participants) | 16 | 11
  36 Hours | 0 (0.11) | 0.1 (0.1)
  42 Hours: number analyzed (Participants) | 16 | 12
  42 Hours | 0 (0.11) | 0.1 (0.09)
  48 Hours: number analyzed (Participants) | 15 | 13
  48 Hours | 0 (0.12) | 0.1 (0.1)
  54 Hours: number analyzed (Participants) | 13 | 10
  54 Hours | 0 (0.13) | 0.1 (0.09)
  60 Hours: number analyzed (Participants) | 13 | 11
  60 Hours | 0 (0.14) | 0.1 (0.08)
  66 Hours: number analyzed (Participants) | 15 | 8
  66 Hours | 0.1 (0.16) | 0 (0.07)
  72 Hours: number analyzed (Participants) | 16 | 10
  72 Hours | 0 (0.13) | 0 (0.16)
  78 Hours: number analyzed (Participants) | 12 | 8
  78 Hours | 0 (0.13) | 0.1 (0.11)
  84 Hours: number analyzed (Participants) | 13 | 9
  84 Hours | 0.1 (0.12) | 0.1 (0.09)
  90 Hours: number analyzed (Participants) | 11 | 9
  90 Hours | 0 (0.14) | 0.1 (0.1)
  96 Hours: number analyzed (Participants) | 12 | 8
  96 Hours | 0 (0.16) | 0.1 (0.14)
  102 Hours: number analyzed (Participants) | 10 | 4
  102 Hours | 0 (0.12) | 0 (0.11)
  108 Hours: number analyzed (Participants) | 12 | 7
  108 Hours | 0 (0.11) | 0.1 (0.16)
  114 Hours: number analyzed (Participants) | 9 | 5
  114 Hours | 0 (0.12) | -0.0 (0.12)
  120 Hours: number analyzed (Participants) | 8 | 5
  120 Hours | -0.0 (0.12) | 0 (0.17)

8. Secondary Outcome: Change From Baseline in Base Excess by Hour
Time Frame: Baseline and up to 120 hours post CRRT treatment initiation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
mmol/L
  6 Hours: number analyzed (Participants) | 12 | 13
  6 Hours | 0.4 (6.92) | 1.1 (4.72)
  12 Hours: number analyzed (Participants) | 13 | 15
  12 Hours | -1.3 (5.06) | 1.7 (4.75)
  18 Hours: number analyzed (Participants) | 15 | 15
  18 Hours | 0.3 (7.28) | 1.1 (6.08)
  24 Hours: number analyzed (Participants) | 16 | 14
  24 Hours | 2.4 (6.65) | 0.6 (6.15)
  30 Hours: number analyzed (Participants) | 14 | 10
  30 Hours | 1.3 (5.64) | 1.7 (5.91)
  36 Hours: number analyzed (Participants) | 16 | 11
  36 Hours | 3 (7.36) | 0.9 (5.74)
  42 Hours: number analyzed (Participants) | 16 | 12
  42 Hours | 2.8 (7.41) | 2.1 (6.09)
  48 Hours: number analyzed (Participants) | 15 | 13
  48 Hours | 2.4 (6.87) | 1.9 (5.67)
  54 Hours: number analyzed (Participants) | 13 | 10
  54 Hours | 1.3 (6.99) | 0.4 (5.78)
  60 Hours: number analyzed (Participants) | 13 | 11
  60 Hours | 3.7 (7.57) | 1.2 (7.26)
  66 Hours: number analyzed (Participants) | 15 | 8
  66 Hours | 3.2 (8.43) | 2.1 (5.2)
  72 Hours: number analyzed (Participants) | 16 | 10
  72 Hours | 3.6 (7.5) | -2.1 (12.94)
  78 Hours: number analyzed (Participants) | 12 | 8
  78 Hours | 2.5 (5.77) | 4 (5.98)
  84 Hours: number analyzed (Participants) | 13 | 9
  84 Hours | 4 (6.61) | 3.7 (5.27)
  90 Hours: number analyzed (Participants) | 11 | 8
  90 Hours | 3 (5.98) | 3.1 (5.53)
  96 Hours: number analyzed (Participants) | 12 | 8
  96 Hours | 3.5 (7.29) | 2.2 (5.91)
  102 Hours: number analyzed (Participants) | 10 | 4
  102 Hours | 1.6 (5.56) | -1.0 (9.04)
  108 Hours: number analyzed (Participants) | 12 | 7
  108 Hours | 3.5 (5.95) | 0.8 (9.34)
  114 Hours: number analyzed (Participants) | 9 | 5
  114 Hours | 2.7 (5.72) | -2.8 (9.47)
  120 Hours: number analyzed (Participants) | 8 | 5
  120 Hours | 2.8 (7.23) | -2.0 (8.94)

9. Secondary Outcome: Change From Baseline in Blood Total Calcium Concentration by Hour
Time Frame: Baseline and up to 120 hours post CRRT treatment initiation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
mmol/L
  1 Hour: number analyzed (Participants) | 13 | 12
  1 Hour | -0.0 (0.12) | -0.0 (0.13)
  6 Hours: number analyzed (Participants) | 16 | 16
  6 Hours | 0.1 (0.21) | -0.0 (0.14)
  12 Hours: number analyzed (Participants) | 15 | 17
  12 Hours | 0.2 (0.27) | -0.0 (0.19)
  18 Hours: number analyzed (Participants) | 13 | 17
  18 Hours | 0.2 (0.25) | -0.0 (0.22)
  24 Hours: number analyzed (Participants) | 14 | 16
  24 Hours | 0.3 (0.24) | -0.1 (0.31)
  30 Hours: number analyzed (Participants) | 13 | 14
  30 Hours | 0.3 (0.22) | -0.0 (0.22)
  36 Hours: number analyzed (Participants) | 15 | 15
  36 Hours | 0.3 (0.24) | -0.1 (0.24)
  42 Hours: number analyzed (Participants) | 14 | 13
  42 Hours | 0.3 (0.28) | -0.1 (0.22)
  48 Hours: number analyzed (Participants) | 14 | 13
  48 Hours | 0.3 (0.26) | -0.1 (0.27)
  54 Hours: number analyzed (Participants) | 15 | 12
  54 Hours | 0.3 (0.24) | -0.1 (0.25)
  60 Hours: number analyzed (Participants) | 14 | 12
  60 Hours | 0.3 (0.24) | -0.1 (0.24)
  66 Hours: number analyzed (Participants) | 14 | 12
  66 Hours | 0.3 (0.27) | -0.1 (0.26)
  72 Hours: number analyzed (Participants) | 15 | 11
  72 Hours | 0.3 (0.27) | -0.1 (0.26)
  78 Hours: number analyzed (Participants) | 12 | 10
  78 Hours | 0.3 (0.29) | -0.1 (0.24)
  84 Hours: number analyzed (Participants) | 12 | 9
  84 Hours | 0.3 (0.33) | -0.2 (0.27)
  90 Hours: number analyzed (Participants) | 11 | 10
  90 Hours | 0.3 (0.35) | -0.1 (0.27)
  96 Hours: number analyzed (Participants) | 11 | 9
  96 Hours | 0.2 (0.27) | -0.2 (0.27)
  102 Hours: number analyzed (Participants) | 11 | 7
  102 Hours | 0.2 (0.27) | -0.1 (0.29)
  108 Hours: number analyzed (Participants) | 11 | 7
  108 Hours | 0.3 (0.35) | -0.1 (0.29)
  114 Hours: number analyzed (Participants) | 9 | 7
  114 Hours | 0.2 (0.27) | -0.2 (0.25)
  120 Hours: number analyzed (Participants) | 6 | 6
  120 Hours | 0.4 (0.2) | -0.1 (0.24)

10. Secondary Outcome: Change From Baseline in Serum Sodium by Hour
Time Frame: Baseline and up to 120 hours post CRRT treatment initiation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
mmol/L
  6 Hours: number analyzed (Participants) | 17 | 16
  6 Hours | -1.1 (2.89) | 0.4 (1.89)
  12 Hours: number analyzed (Participants) | 16 | 17
  12 Hours | -1.6 (2.06) | -0.1 (3.01)
  18 Hours: number analyzed (Participants) | 14 | 17
  18 Hours | -1.7 (2.13) | 0.5 (3.39)
  24 Hours: number analyzed (Participants) | 15 | 16
  24 Hours | -1.7 (4.19) | 0.4 (4.35)
  30 Hours: number analyzed (Participants) | 14 | 14
  30 Hours | -1.9 (4.03) | 0.4 (4.83)
  36 Hours: number analyzed (Participants) | 16 | 15
  36 Hours | -1.1 (5.13) | -0.3 (5.08)
  42 Hours: number analyzed (Participants) | 15 | 13
  42 Hours | -0.7 (5.15) | -0.4 (5.04)
  48 Hours: number analyzed (Participants) | 15 | 13
  48 Hours | -1.5 (5.74) | 1.2 (4.47)
  54 Hours: number analyzed (Participants) | 16 | 12
  54 Hours | -1.3 (6.29) | 0.5 (4.95)
  60 Hours: number analyzed (Participants) | 15 | 12
  60 Hours | -1.3 (5.86) | 1 (4.99)
  66 Hours: number analyzed (Participants) | 15 | 12
  66 Hours | -0.7 (6.1) | 0.3 (4.11)
  72 Hours: number analyzed (Participants) | 16 | 11
  72 Hours | -0.8 (5.62) | 2.5 (4.61)
  78 Hours: number analyzed (Participants) | 13 | 10
  78 Hours | -1.8 (5.21) | 2.6 (4.06)
  84 Hours: number analyzed (Participants) | 13 | 9
  84 Hours | -2.2 (4.95) | 1.7 (4.87)
  90 Hours: number analyzed (Participants) | 12 | 10
  90 Hours | -1.8 (4.17) | 2.2 (4.47)
  96 Hours: number analyzed (Participants) | 12 | 9
  96 Hours | -2.0 (4.51) | 2.3 (3.24)
  102 Hours: number analyzed (Participants) | 12 | 7
  102 Hours | -1.8 (4.9) | 1.1 (3.53)
  108 Hours: number analyzed (Participants) | 12 | 7
  108 Hours | -2.4 (4.36) | 0.7 (3.73)
  114 Hours: number analyzed (Participants) | 10 | 7
  114 Hours | -2.8 (4.78) | 1.4 (4.12)
  120 Hours: number analyzed (Participants) | 7 | 7
  120 Hours | -3.7 (4.39) | 1 (5.16)

11. Secondary Outcome: Change From Baseline in Serum Anion Gap by Hour
Time Frame: Baseline and up to 120 hours post CRRT treatment initiation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
mmol/L
  6 Hours: number analyzed (Participants) | 17 | 16
  6 Hours | 0.6 (3.08) | -2.3 (2.27)
  12 Hours: number analyzed (Participants) | 16 | 17
  12 Hours | 0.6 (2.45) | -3.5 (3.1)
  18 Hours: number analyzed (Participants) | 15 | 17
  18 Hours | 0.2 (2.96) | -2.2 (4.72)
  24 Hours: number analyzed (Participants) | 15 | 16
  24 Hours | -0.5 (3.07) | -2.9 (3.24)
  30 Hours: number analyzed (Participants) | 14 | 14
  30 Hours | 1.6 (3.08) | -3.6 (3.55)
  36 Hours: number analyzed (Participants) | 16 | 15
  36 Hours | 0.5 (3.41) | -4 (2.73)
  42 Hours: number analyzed (Participants) | 15 | 13
  42 Hours | 0.7 (3.33) | -3.5 (2.9)
  48 Hours: number analyzed (Participants) | 15 | 13
  48 Hours | 0.7 (3.7) | -2.8 (3.21)
  54 Hours: number analyzed (Participants) | 16 | 12
  54 Hours | 0.3 (3.47) | -3.2 (3.27)
  60 Hours: number analyzed (Participants) | 15 | 12
  60 Hours | 0.4 (3.58) | -2.3 (3.67)
  66 Hours: number analyzed (Participants) | 15 | 12
  66 Hours | 1.1 (4) | -3.2 (4.37)
  72 Hours: number analyzed (Participants) | 16 | 11
  72 Hours | 1 (4.37) | 0 (5.93)
  78 Hours: number analyzed (Participants) | 13 | 10
  78 Hours | 0.7 (2.39) | -2.0 (3.4)
  84 Hours: number analyzed (Participants) | 13 | 9
  84 Hours | 0.8 (2.74) | -3.0 (3.91)
  90 Hours: number analyzed (Participants) | 12 | 10
  90 Hours | 0.8 (3.59) | -2.1 (3.54)
  96 Hours: number analyzed (Participants) | 12 | 9
  96 Hours | 1.6 (2.35) | -1.7 (4.21)
  102 Hours: number analyzed (Participants) | 12 | 7
  102 Hours | 1.5 (2.54) | -1.7 (5.15)
  108 Hours: number analyzed (Participants) | 12 | 7
  108 Hours | 0.8 (2.67) | 0.6 (5.44)
  114 Hours: number analyzed (Participants) | 10 | 7
  114 Hours | 1 (2.71) | 0.7 (8.64)
  120 Hours: number analyzed (Participants) | 7 | 6
  120 Hours | -0.3 (2.06) | -1.2 (7.03)

12. Secondary Outcome: Change From Baseline in Serum Magnesium by Hour
Time Frame: Baseline and up to 120 hours post CRRT treatment initiation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
mmol/L
  6 Hours: number analyzed (Participants) | 15 | 16
  6 Hours | -0.1 (0.12) | 0 (0.14)
  12 Hours: number analyzed (Participants) | 14 | 17
  12 Hours | -0.1 (0.14) | -0.0 (0.14)
  18 Hours: number analyzed (Participants) | 12 | 17
  18 Hours | -0.1 (0.19) | 0 (0.14)
  24 Hours: number analyzed (Participants) | 13 | 16
  24 Hours | -0.2 (0.2) | -0.0 (0.16)
  30 Hours: number analyzed (Participants) | 11 | 13
  30 Hours | -0.1 (0.23) | 0 (0.17)
  36 Hours: number analyzed (Participants) | 14 | 15
  36 Hours | -0.1 (0.22) | 0 (0.19)
  42 Hours: number analyzed (Participants) | 13 | 13
  42 Hours | -0.2 (0.23) | 0 (0.2)
  48 Hours: number analyzed (Participants) | 12 | 13
  48 Hours | -0.2 (0.25) | 0.1 (0.16)
  54 Hours: number analyzed (Participants) | 14 | 12
  54 Hours | -0.2 (0.21) | 0 (0.2)
  60 Hours: number analyzed (Participants) | 13 | 12
  60 Hours | -0.1 (0.23) | 0 (0.2)
  66 Hours: number analyzed (Participants) | 13 | 12
  66 Hours | -0.1 (0.24) | 0 (0.18)
  72 Hours: number analyzed (Participants) | 13 | 11
  72 Hours | -0.1 (0.22) | 0.1 (0.2)
  78 Hours: number analyzed (Participants) | 10 | 10
  78 Hours | -0.2 (0.21) | 0.1 (0.16)
  84 Hours: number analyzed (Participants) | 11 | 9
  84 Hours | -0.2 (0.22) | 0 (0.18)
  90 Hours: number analyzed (Participants) | 10 | 10
  90 Hours | -0.2 (0.27) | 0.1 (0.21)
  96 Hours: number analyzed (Participants) | 10 | 9
  96 Hours | -0.2 (0.24) | 0.1 (0.18)
  102 Hours: number analyzed (Participants) | 10 | 7
  102 Hours | -0.2 (0.23) | 0.1 (0.2)
  108 Hours: number analyzed (Participants) | 10 | 7
  108 Hours | -0.2 (0.28) | 0.1 (0.2)
  114 Hours: number analyzed (Participants) | 8 | 7
  114 Hours | -0.1 (0.27) | 0.1 (0.23)
  120 Hours: number analyzed (Participants) | 6 | 6
  120 Hours | -0.2 (0.28) | 0 (0.21)

13. Secondary Outcome: Change From Baseline in Serum Phosphate by Hour
Time Frame: Baseline and up to 120 hours post CRRT treatment initiation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
mmol/L
  6 Hours: number analyzed (Participants) | 15 | 15
  6 Hours | -0.3 (0.33) | -0.4 (0.29)
  12 Hours: number analyzed (Participants) | 14 | 16
  12 Hours | -0.3 (0.51) | -0.4 (0.32)
  18 Hours: number analyzed (Participants) | 11 | 16
  18 Hours | -0.5 (0.7) | -0.4 (0.41)
  24 Hours: number analyzed (Participants) | 13 | 15
  24 Hours | -0.7 (0.74) | -0.4 (0.36)
  30 Hours: number analyzed (Participants) | 12 | 13
  30 Hours | -0.6 (0.7) | -0.5 (0.35)
  36 Hours: number analyzed (Participants) | 14 | 14
  36 Hours | -0.7 (0.78) | -0.4 (0.32)
  42 Hours: number analyzed (Participants) | 14 | 12
  42 Hours | -0.8 (0.82) | -0.5 (0.32)
  48 Hours: number analyzed (Participants) | 13 | 12
  48 Hours | -0.9 (0.87) | -0.4 (0.33)
  54 Hours: number analyzed (Participants) | 14 | 11
  54 Hours | -0.8 (0.86) | -0.4 (0.43)
  60 Hours: number analyzed (Participants) | 13 | 11
  60 Hours | -0.9 (0.93) | -0.4 (0.41)
  66 Hours: number analyzed (Participants) | 12 | 11
  66 Hours | -0.8 (0.89) | -0.4 (0.52)
  72 Hours: number analyzed (Participants) | 13 | 10
  72 Hours | -0.8 (0.88) | -0.2 (0.74)
  78 Hours: number analyzed (Participants) | 10 | 9
  78 Hours | -0.8 (0.86) | -0.4 (0.55)
  84 Hours: number analyzed (Participants) | 10 | 8
  84 Hours | -0.8 (0.84) | -0.4 (0.48)
  90 Hours: number analyzed (Participants) | 10 | 9
  90 Hours | -0.8 (0.84) | -0.3 (0.71)
  96 Hours: number analyzed (Participants) | 10 | 8
  96 Hours | -0.8 (0.92) | -0.5 (0.6)
  102 Hours: number analyzed (Participants) | 10 | 7
  102 Hours | -0.7 (0.85) | -0.4 (0.63)
  108 Hours: number analyzed (Participants) | 10 | 6
  108 Hours | -0.8 (0.84) | -0.4 (0.76)
  114 Hours: number analyzed (Participants) | 8 | 5
  114 Hours | -0.9 (0.91) | 0.2 (0.77)
  120 Hours: number analyzed (Participants) | 7 | 5
  120 Hours | -0.8 (1.02) | -0.2 (0.86)

14. Secondary Outcome: Change From Baseline in Serum Potassium by Hour
Time Frame: Baseline and up to 120 hours post CRRT treatment initiation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
mmol/L
  6 Hours: number analyzed (Participants) | 17 | 16
  6 Hours | -0.4 (0.62) | -0.1 (0.56)
  12 Hours: number analyzed (Participants) | 16 | 17
  12 Hours | -0.4 (0.66) | -0.1 (0.51)
  18 Hours: number analyzed (Participants) | 14 | 17
  18 Hours | -0.7 (0.68) | -0.1 (0.43)
  24 Hours: number analyzed (Participants) | 15 | 16
  24 Hours | -0.9 (0.75) | -0.2 (0.49)
  30 Hours: number analyzed (Participants) | 14 | 14
  30 Hours | -0.9 (0.7) | -0.1 (0.67)
  36 Hours: number analyzed (Participants) | 16 | 15
  36 Hours | -1.0 (0.81) | -0.0 (0.69)
  42 Hours: number analyzed (Participants) | 15 | 13
  42 Hours | -1.0 (0.68) | -0.0 (0.58)
  48 Hours: number analyzed (Participants) | 15 | 13
  48 Hours | -1.0 (0.62) | -0.0 (0.54)
  54 Hours: number analyzed (Participants) | 16 | 12
  54 Hours | -1.2 (0.61) | 0.1 (0.65)
  60 Hours: number analyzed (Participants) | 15 | 12
  60 Hours | -1.2 (0.76) | 0.1 (0.54)
  66 Hours: number analyzed (Participants) | 15 | 12
  66 Hours | -1.2 (0.81) | 0.3 (0.58)
  72 Hours: number analyzed (Participants) | 16 | 11
  72 Hours | -1.2 (0.69) | 0.2 (0.83)
  78 Hours: number analyzed (Participants) | 13 | 10
  78 Hours | -1.2 (0.75) | 0.1 (0.68)
  84 Hours: number analyzed (Participants) | 13 | 9
  84 Hours | -1.3 (0.77) | 0.2 (0.65)
  90 Hours: number analyzed (Participants) | 12 | 10
  90 Hours | -1.4 (0.71) | 0.2 (0.75)
  96 Hours: number analyzed (Participants) | 12 | 9
  96 Hours | -1.1 (0.85) | 0.2 (0.82)
  102 Hours: number analyzed (Participants) | 12 | 7
  102 Hours | -1.2 (0.72) | 0 (0.73)
  108 Hours: number analyzed (Participants) | 12 | 7
  108 Hours | -1.2 (0.76) | 0.1 (0.86)
  114 Hours: number analyzed (Participants) | 10 | 7
  114 Hours | -1.5 (0.8) | 0.2 (0.85)
  120 Hours: number analyzed (Participants) | 7 | 7
  120 Hours | -1.1 (0.63) | 0.1 (0.75)

15. Secondary Outcome: Change From Baseline in Serum Chloride by Hour
Time Frame: Baseline and up to 120 hours post CRRT treatment initiation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
mmol/L
  6 Hours: number analyzed (Participants) | 17 | 16
  6 Hours | -1.9 (4.12) | 0.6 (3.1)
  12 Hours: number analyzed (Participants) | 16 | 17
  12 Hours | -3.4 (4.23) | 0.9 (3.44)
  18 Hours: number analyzed (Participants) | 14 | 17
  18 Hours | -3.9 (5.67) | 0.8 (3.52)
  24 Hours: number analyzed (Participants) | 15 | 16
  24 Hours | -3.9 (6.58) | 1.3 (5.04)
  30 Hours: number analyzed (Participants) | 14 | 14
  30 Hours | -5.5 (6.84) | 1.1 (4.59)
  36 Hours: number analyzed (Participants) | 16 | 15
  36 Hours | -5.0 (6.73) | 0.6 (4.44)
  42 Hours: number analyzed (Participants) | 15 | 13
  42 Hours | -4.9 (7.31) | 0.5 (4.5)
  48 Hours: number analyzed (Participants) | 15 | 13
  48 Hours | -5.1 (7.35) | 1.3 (4.44)
  54 Hours: number analyzed (Participants) | 16 | 12
  54 Hours | -5.4 (7.39) | 0.9 (4.91)
  60 Hours: number analyzed (Participants) | 15 | 12
  60 Hours | -5.9 (7.68) | 1 (4.79)
  66 Hours: number analyzed (Participants) | 15 | 12
  66 Hours | -5.3 (7.82) | 1 (4.94)
  72 Hours: number analyzed (Participants) | 16 | 11
  72 Hours | -5.6 (7.61) | 1.7 (4.38)
  78 Hours: number analyzed (Participants) | 13 | 10
  78 Hours | -5.5 (7.4) | 2.4 (4.45)
  84 Hours: number analyzed (Participants) | 13 | 9
  84 Hours | -5.8 (6.76) | 2.1 (5.33)
  90 Hours: number analyzed (Participants) | 12 | 10
  90 Hours | -5.9 (7.68) | 2.3 (5.1)
  96 Hours: number analyzed (Participants) | 12 | 9
  96 Hours | -6.2 (7.69) | 2.4 (4.64)
  102 Hours: number analyzed (Participants) | 12 | 7
  102 Hours | -6.0 (7.51) | 2.6 (6.02)
  108 Hours: number analyzed (Participants) | 12 | 7
  108 Hours | -5.9 (7.88) | 1.3 (4.42)
  114 Hours: number analyzed (Participants) | 10 | 7
  114 Hours | -7.7 (8.63) | 1.1 (5.96)
  120 Hours: number analyzed (Participants) | 7 | 7
  120 Hours | -8.1 (6.28) | 1 (5.89)

16. Secondary Outcome: Number of Participants With Bleeding Events
Time Frame: Up to 120 hours post CRRT treatment initiation
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
Participants
  0 Bleeding Events | 16 | 13
  1 Bleeding Events | 1 | 3
  2 Bleeding Events | 0 | 0
  4 Bleeding Events | 0 | 1

17. Secondary Outcome: Number of Participants by Number of Blood Transfusions
Time Frame: Up to 120 hours post CRRT treatment initiation
Population: FAS
Measure: Number; unit: participants
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
participants
  3 Transfusions | 1 | 2
  27 Transfusions | 0 | 1

18. Secondary Outcome: Number of Participants Reporting Any Baxter Device/Product Related Adverse Events (Serious and Non-Serious)
Time Frame: Up to 30 days post study CRRT treatment completion
Population: FAS
Measure: Number; unit: Events
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
Events | 0 | 1

19. Secondary Outcome: Change From Baseline in Blood Pressure at Last Visit
Time Frame: Baseline and up to 120 hours post CRRT treatment initiation
Population: FAS
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
mmHg
  Systolic | 1.9 (25.37) | -6.4 (30.99)
  Diastolic | -2.8 (12.29) | 2.8 (21.19)

20. Secondary Outcome: Change From Baseline in Respiratory Rate at Last Visit
Time Frame: Baseline and up to 120 hours post CRRT treatment initiation
Population: FAS
Measure: Mean (Standard Deviation); unit: breaths/Min
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
breaths/Min | -2.1 (5.42) | -1.1 (7.64)

21. Secondary Outcome: Change From Baseline in Temperature at Last Visit
Time Frame: Baseline and up to 120 hours post CRRT treatment initiation
Population: FAS
Measure: Mean (Standard Deviation); unit: degree celsius
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
degree celsius | 0.2 (0.69) | -0.1 (1.12)

22. Secondary Outcome: Change From Baseline in Pulse at Last Visit
Time Frame: Baseline and up to 120 hours post CRRT treatment initiation
Population: FAS
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
beats/min | 2.1 (24.66) | 3.2 (16.52)

23. Secondary Outcome: Change From Baseline in Total Calcium/iCa Ratio by Hour
Time Frame: Baseline and up to 120 hours post CRRT treatment initiation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
ratio
  1 Hour: number analyzed (Participants) | 14 | 12
  1 Hour | 0.2 (0.25) | -0.1 (0.12)
  6 Hours: number analyzed (Participants) | 16 | 15
  6 Hours | 0.2 (0.17) | -0.1 (0.12)
  12 Hours: number analyzed (Participants) | 14 | 15
  12 Hours | 0.2 (0.18) | -0.1 (0.12)
  18 Hours: number analyzed (Participants) | 16 | 15
  18 Hours | 0.2 (0.13) | -0.1 (0.1)
  24 Hours: number analyzed (Participants) | 14 | 14
  24 Hours | 0.3 (0.25) | -0.1 (0.08)
  30 Hours: number analyzed (Participants) | 15 | 13
  30 Hours | 0.2 (0.16) | -0.1 (0.09)
  36 Hours: number analyzed (Participants) | 15 | 12
  36 Hours | 0.2 (0.14) | -0.1 (0.08)
  42 Hours: number analyzed (Participants) | 14 | 13
  42 Hours | 0.3 (0.21) | -0.1 (0.08)
  48 Hours: number analyzed (Participants) | 14 | 13
  48 Hours | 0.2 (0.2) | -0.1 (0.07)
  54 Hours: number analyzed (Participants) | 15 | 11
  54 Hours | 0.2 (0.18) | -0.1 (0.1)
  60 Hours: number analyzed (Participants) | 14 | 10
  60 Hours | 0.2 (0.16) | -0.1 (0.09)
  66 Hours: number analyzed (Participants) | 14 | 11
  66 Hours | 0.2 (0.19) | -0.1 (0.09)
  72 Hours: number analyzed (Participants) | 15 | 10
  72 Hours | 0.2 (0.16) | -0.1 (0.1)
  78 Hours: number analyzed (Participants) | 12 | 9
  78 Hours | 0.2 (0.23) | -0.1 (0.13)
  84 Hours: number analyzed (Participants) | 12 | 9
  84 Hours | 0.2 (0.18) | -0.1 (0.09)
  90 Hours: number analyzed (Participants) | 11 | 8
  90 Hours | 0.2 (0.18) | -0.1 (0.11)
  96 Hours: number analyzed (Participants) | 11 | 8
  96 Hours | 0.2 (0.2) | -0.1 (0.11)
  102 Hours: number analyzed (Participants) | 11 | 6
  102 Hours | 0.2 (0.2) | -0.1 (0.11)
  108 Hours: number analyzed (Participants) | 11 | 6
  108 Hours | 0.2 (0.19) | -0.1 (0.14)
  114 Hours: number analyzed (Participants) | 9 | 6
  114 Hours | 0.1 (0.17) | -0.1 (0.11)
  120 Hours: number analyzed (Participants) | 6 | 4
  120 Hours | 0.2 (0.14) | -0.1 (0.09)

24. Secondary Outcome: Number of Bleeding Events by Location
Time Frame: Up to 120 hours post CRRT treatment initiation
Population: FAS
Measure: Number; unit: Events
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
Events
  Gastrointestinal | 1 | 4
  M150 filter | 0 | 1
  ostomy and rectum | 0 | 1
  upper Gastrointestinal tract | 0 | 1

25. Secondary Outcome: Duration of Bleeding Events
Time Frame: Up to 120 hours post CRRT treatment initiation
Population: FAS
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
Number analyzed (Participants) | 17 | 17
Hours | 0 (0) | 14.4 (12.71)

ADVERSE EVENTS:
Time Frame: Up to 120 hours post CRRT treatment initiation
Arm/Group | Prismocitrate 18 | No Systemic Anticoagulation
All-Cause Mortality (participants affected / at risk) | 8/17 | 9/17
Serious Adverse Events (participants affected / at risk) | 10/17 | 10/17
Other Adverse Events (participants affected / at risk) | 13/17 | 14/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prismocitrate 18 (N=17) | No Systemic Anticoagulation (N=17)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (3)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cardiac death (General disorders) | 0 (0) | 2 (2)
Death (General disorders) | 1 (1) | 0 (0)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 4 (5) | 2 (2)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood lactic acid increased (Investigations) | 0 (0) | 1 (1)
Blood pH decreased (Investigations) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prismocitrate 18 (N=17) | No Systemic Anticoagulation (N=17)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 6 (6) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hypophosphatasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eye complication associated with device (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Therapeutic response decreased (General disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood bicarbonate decreased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood chloride decreased (Investigations) | 0 (0) | 1 (1)
Blood lactic acid increased (Investigations) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (2)
Hepatic enzyme abnormal (Investigations) | 0 (0) | 1 (1)
PCO2 decreased (Investigations) | 0 (0) | 1 (1)
Radial pulse abnormal (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Anuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Axillary vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
The study was terminated as it was proven to be extremely difficult to enroll patients. The study termination decision was unrelated to safety or efficacy. Given the early termination, this study was not powered to show statistically significant changes in efficacy endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reserves the right of prior review and approval of data from this study relative to the potential release of proprietary information to any publication or for any presentation.

DOCUMENTS (2):
  • Study Protocol (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT02860130/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT02860130/SAP_001.pdf